CLINICAL TRIAL: NCT02634346
Title: A Phase 3 Study to Determine the Antipsychotic Efficacy and Safety of ALKS 3831 in Adult Subjects With Acute Exacerbation of Schizophrenia
Brief Title: A Study of ALKS 3831 in Adults With Acute Exacerbation of Schizophrenia (the ENLIGHTEN-1 Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALKS-3831-A305
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia
Keywords: Alkermes; ALKS 3831; Samidorphan; Schizophrenia; Acute Exacerbation of Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALKS 3831 (Experimental): Administered as a coated bilayer tablet
  Interventions: Drug: ALK3831
- Olanzapine (Active Comparator): Administered as a coated bilayer tablet
  Interventions: Drug: Olanzapine
- Placebo (Placebo Comparator): Administered as a coated bilayer tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALK3831 — Daily dosing
  Arms: ALKS 3831
Drug: Olanzapine — Daily dosing
  Arms: Olanzapine
Drug: Placebo — Daily dosing
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of ALKS 3831 in adult subjects with acute exacerbation of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) of 18.0 - 40.0 kg/m^2
* Meets criteria for the diagnosis of schizophrenia
* Resides in a stable living situation when not hospitalized
* Is willing and able to provide government-issued identification
* Additional criteria may apply

Exclusion Criteria:

* Has had a psychiatric hospitalization for more than 30 days during the 90 days before screening
* Subject initiated first antipsychotic treatment within the past 12 months, or <1 year has elapsed since the initial onset of active-phase of schizophrenia symptoms
* Subject poses a current suicide risk
* Subject has a history of treatment resistance
* Subject has a history of poor or inadequate response to treatment with olanzapine
* Subject requires or has had electroconvulsive therapy (ECT) treatment in the 2-month period prior to screening
* Subject has a diagnosis of moderate or severe alcohol or drug use disorder
* Subject has a positive urine drug screen for opioids, amphetamine/methamphetamine, phencyclidine, or cocaine at screening
* Additional criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David McDonnell, MD, Study Director — Alkermes, Inc.
Locations (31):
- United States (16):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Springdale, Arkansas
  - Alkermes Investigational Site, Culver City, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Lemon Grove, California
  - Alkermes Investigational Site, Long Beach, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, North Miami, Florida
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Marlton, New Jersey
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Dallas, Texas
- Bulgaria (7):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Kazanlak
  - Alkermes Investigational Site, Lovech
  - Alkermes Investigational Site, Novi Iskar
  - Alkermes Investigational Site, Plovdiv
  - Alkermes Investigational Site, Veliko Tarnovo
  - Alkermes Investigational Site, Vratsa
- Serbia (3):
  - Alkermes Investigational Site, Belgrade
  - Alkermes Investigational Site, Kragujevac
  - Alkermes Investigational Site, Novi Kneževac
- Ukraine (5):
  - Alkermes Investigational Site, Cherkasy
  - Alkermes Investigational Site, Kherson
  - Alkermes Investigational Site, Kiev
  - Alkermes Investigational Site, Lviv
  - Alkermes Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Potkin SG, Kunovac J, Silverman BL, Simmons A, Jiang Y, DiPetrillo L, McDonnell D. Efficacy and Safety of a Combination of Olanzapine and Samidorphan in Adult Patients With an Acute Exacerbation of Schizophrenia: Outcomes From the Randomized, Phase 3 ENLIGHTEN-1 Study. J Clin Psychiatry. 2020 Mar 3;81(2):19m12769. doi: 10.4088/JCP.19m12769. PMID 32141723

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Disposition is shown for the safety population - subjects who were randomized and received at least 1 dose of study drug. 1 subject in the placebo group and 1 subject in the olanzapine-only group were randomized but not treated, and thus were not included in the safety population.
Groups:
- ALKS 3831: Olanzapine + samidorphan; administered as a coated bilayer tablet
  ALK3831: Daily dosing
Period: Overall Study
Arm/Group | ALKS 3831 | Olanzapine | Placebo
Started | 134 | 133 | 134
Completed | 122 | 119 | 111
Not Completed | 12 | 14 | 23
Not completed — Withdrawal by Subject | 8 | 9 | 8
Not completed — Adverse Event | 2 | 2 | 7
Not completed — Lack of Efficacy | 1 | 2 | 8
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Disposition is shown for all subjects randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALKS 3831 | Olanzapine | Placebo | Total
Number analyzed (Participants) | 134 | 133 | 134 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (12.55) | 41.5 (10.89) | 41.1 (10.59) | 41.1 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 52 | 56 | 157
  Male | 85 | 81 | 78 | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 4 | 13
  Not Hispanic or Latino | 132 | 126 | 130 | 388
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 42 | 33 | 38 | 113
  White | 87 | 99 | 91 | 277
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 55 | 50 | 49 | 154
  Ukraine | 24 | 26 | 29 | 79
  Bulgaria | 44 | 38 | 45 | 127
  Serbia | 11 | 19 | 11 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 4
Description: This scale consists of symptom constructs (7 positive, 7 negative, 16 general psychopathology), each to be rated on a 7-point Likert-type scale of severity with 1 being absent to 7 being extreme. Minimum scores (best outcome) equals 30 (total scale); maximum scores (worst outcome) equals 210 (total scale). Change is calculated between the baseline visit and Week 4.
Time Frame: 4 weeks
Population: Subjects that received at least 1 dose of study drug and had at least 1 post-baseline PANSS assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ALKS 3831 | Olanzapine | Placebo
Number analyzed (Participants) | 132 | 132 | 133
units on a scale | -23.9 (1.28) | -22.8 (1.29) | -17.5 (1.32)
Statistical Analysis 1: Comparison: ALKS 3831 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mixed model for repeated measures is based on observed data without imputation of missing data; Least square mean difference = -6.4, 95% CI 2-sided [-10.0 to -2.8], Standard Error of Mean 1.83
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mixed model for repeated measures is based on observed data without imputation of missing data; Least square mean difference = -5.3, 95% CI 2-sided [-8.9 to -1.7], Standard Error of Mean 1.84

2. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Severity (CGIS) Score at Week 4
Description: The CGI-S is a 7-point scale that requires the clinician to assess how mentally ill the patient is in a specific point in time. Results indicate participants evaluated at one of the following categories: "1: normal, not at all ill"; "2: borderline mentally ill"; "3: mildly ill"; "4: moderately ill"; "5: markedly ill"; "6: severely ill"; and "7: among the most extremely ill patients". Results indicate a change in CGI-S score from baseline to Week 4 based on the observed data. Change is calculated between the baseline visit and Week 4.
Time Frame: 4 weeks
Population: Subjects who received at least 1 dose of study drug and had at least 1 post-baseline PANSS assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ALKS 3831 | Olanzapine | Placebo
Number analyzed (Participants) | 132 | 132 | 133
units on a scale | -1.21 (0.082) | -1.27 (0.083) | -0.84 (0.085)
Statistical Analysis 1: Comparison: ALKS 3831 vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mixed model for repeated measures is based on observed data without imputation of missing data; Least square mean difference = -0.38, 95% CI 2-sided [-0.61 to -0.14], Standard Error of Mean 0.118
Statistical Analysis 2: Comparison: Olanzapine vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mixed model for repeated measures is based on observed data without imputation of missing data; Least square mean difference = -0.44, 95% CI 2-sided [-0.67 to -0.20], Standard Error of Mean 0.118

3. Secondary Outcome: Incidence of Adverse Events
Time Frame: Approximately 4 weeks
Population: Number of subjects who received study drug and had a treatment-emergent adverse event
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 3831 | Olanzapine | Placebo
Number analyzed (Participants) | 134 | 133 | 134
Participants | 73 | 73 | 60

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are presented for the double-blind treatment period (4 weeks).
Description: The safety population includes all subjects who received at least 1 dose of study drug.
Arm/Group | ALKS 3831 | Olanzapine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/134 | 1/133 | 0/134
Serious Adverse Events (participants affected / at risk) | 1/134 | 1/133 | 0/134
Other Adverse Events (participants affected / at risk) | 50/134 | 45/133 | 24/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 3831 (N=134) | Olanzapine (N=133) | Placebo (N=134)
Catatonia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 3831 (N=134) | Olanzapine (N=133) | Placebo (N=134)
Weight increased (Investigations) | 25 (25) | 19 (19) | 4 (4)
Somnolence (Nervous system disorders) | 12 (12) | 13 (13) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 10 (10) | 7 (8) | 1 (1)
Anxiety (Psychiatric disorders) | 8 (8) | 7 (7) | 8 (12)
Headache (Nervous system disorders) | 8 (8) | 7 (9) | 4 (7)
Schizophrenia (Psychiatric disorders) | 1 (1) | 2 (2) | 8 (8)

LIMITATIONS AND CAVEATS:
The dose of olanzapine was not fixed and could be titrated during the first 2 weeks of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT02634346/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT02634346/SAP_001.pdf